CLINICAL TRIAL: NCT05434988
Title: Outcome and Quality of Life in Obese Patients Underwent Laparoscopic vs. Open Appendectomy
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Waleed Ghareeb, Lecturer, Suez Canal University
Other Study IDs: 4245/2020
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Obesity; Appendicitis Acute
Keywords: Appendicitis; Obesity; laparoscopic appendectomy
MeSH Terms: conditions — Obesity; Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic appendectomy: The laparoscopic appendectomy group is the group that includes patients who underwent appendectomy using the laparoscopic approach
  Interventions: Procedure: appendectomy
- Open appendectomy: The open appendectomy group is the group that includes patients who underwent appendectomy using laparoscopic approach
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Procedure: appendectomy — Open or Laparoscopic appendectomy procedure is typically performed under general anaesthesia. in the laparoscopic approach, the main principle is the triangulation of instrument ports to visualize and expose the appendix clearly. The first trocar (10 mm) for the optical device is introduced peri-umbilically, followed by two 5 mm trocars, one in the right lower quadrant just above the pubis (to grasp the appendix) and the other in the left iliac fossa (for the (right-handed) surgeon's right hand), assuming the appendix is in its normal anatomic position. The locations of the 5 mm trocars can be changed based on the anatomic position of the appendix as determined before to surgery (for example a subhepatic appendix could lead to placing the trocars as for cholecystectomy)

SUMMARY:
Although obesity is a popular reason for choosing laparoscopic appendectomy (LA) versus open appendectomy (OA), however, the question of whether there is a difference remains. The goal of the present study is to investigate if there is a difference between OA and LA in obese patients. In the present study, Fifty-eight obese patients were diagnosed with acute appendicitis according to Alvarado score at the department of surgery at Suez Canal university hospitals from March 2020 till August 2021were included. The study participants were assigned to two groups, after their approval: LA and OA. The investigators hypothesized that evaluating the Outcome and Quality of life of laparoscopic appendectomy for the obese patients would be a potential step for standardization of the laparoscopic approach for obese patients who are arranged for appendectomy.

DETAILED DESCRIPTION:
Although obesity is a popular reason for choosing laparoscopic appendectomy (LA) versus open appendectomy (OA), however, the question of whether there is a difference remains. The investigators' goal is to investigate if there is a difference between OA and LA in obese patients. Fifty-eight obese patients were diagnosed with acute appendicitis according to Alvarado score at the department of surgery at Suez Canal university hospitals from March 2020 till August 2021were included. The study participants were assigned to two groups, LA and OA. This study aimed to compare LA and OA regarding intraoperative complications, length of hospital stays, post-operative pain, and rate of postoperative complications. Meanwhile, using the SF-36 scoring questionnaire, the quality of life was compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-40 years, with BMI ≥ 30 kg/m2 and diagnosed as acute appendicitis according to Alvarado score i.e., history of right lower quadrant pain or peri-umbilical pain shifting to the right lower quadrant with nausea and/or vomiting, fever of more than 38ºC, right lower quadrant guarding, and tenderness on physical examination and/or leukocytosis above 10,000 cells per ml were included.

Exclusion Criteria:

* The investigators excluded patients with a bleeding tendency., previous lower abdominal surgery, abdominal tuberculosis, mass formation either clinically or by ultrasound, end-stage renal disease (ESRD) patients, and patients who refused to participate in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: obese patients (body mass index >30kg/m2) who were diagnosed with acute appendicitis according to ALVARDO score at the department of surgery at Suez Canal university hospitals
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
The grade of The Clavien-Dindo for postoperative complications | 30 days
  compare the laparoscopic appendectomy vs. Open appendectomy in terms of intraoperative and postoperative complications during the 30 days postoperative (The Clavien-Dindo )
The score for quality of life | 30 days
  the postoperative quality of life has been compared between both groups using SF-36 scoring questionnaire. The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). The higher scores mean better quality of life..

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Hussein, MD, PhD, Study Director — Suez canal University, Faculty of Medicine
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No
All data are available with the principal investigator on reasonable request